CLINICAL TRIAL: NCT04848597
Title: Phase 2, Open-label, Single Center, Prospective Study of Recombinant Humanized Anti-PD-1 Monoclonal Antibody Combined With Nab-paclitaxel and Bevacizumab in the Second-line Treatment of Patients With Cancer of Unknown Primary (CUP)
Brief Title: PD-1 Inhibitor and Nab-paclitaxel and Bevacizumab in CUP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xichun Hu, Director of department of medical oncology, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CUP-002
Record Dates: First submitted 2021-04-14; First posted 2021-04-19 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Cancer of Unknown Primary
MeSH Terms: interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm (Experimental): Recombinant humanized anti-PD-1 monoclonal antibody injection:200mg once every 3 weeks
  Interventions: Drug: Recombinant humanized anti-PD-1 monoclonal antibody injection

INTERVENTIONS:
Drug: Recombinant humanized anti-PD-1 monoclonal antibody injection — 200mg , once every 3 weeks
  Other Names: Albumin Paclitaxel; bevacizumab

SUMMARY:
This trial is a single-center, prospective, single-arm Phase II clinical study. The purpose is to evaluate the efficacy and safety of recombinant humanized anti-PD-1 monoclonal antibody combined with albumin paclitaxel and bevacizumab in the second-line treatment of patients with unknown primary tumors.

DETAILED DESCRIPTION:
Recombinant humanized anti-PD-1 monoclonal antibody combined with albumin paclitaxel and bevacizumab treatment, once every 3 weeks, treatment until disease progression, intolerable adverse reactions, patient death or withdrawal informed agree.After treatment, the patients was followed up every 9 weeks for follow-up treatment and survival.

ELIGIBILITY:
Inclusion Criteria:

1. The histopathologically confirmed metastasis is adenocarcinoma, squamous cell carcinoma, poorly differentiated carcinoma, poorly differentiated malignant tumor or neuroendocrine carcinoma;
2. Patients whose primary lesions cannot be found after standard evaluation prior to treatment: detailed history, physical examination, blood test, chest and pelvic CT, PET/CT (optional), endoscopy of symptomatic sites, and pathological examination;
3. Measurable lesions (RECIST 1.1 criteria);
4. Patients who have progressed after receiving first-line treatment for Carcinoma of Unknown Primary. For example, those who have received paclitaxel or docetaxel in the first-line treatment and progressed more than three months after the end of last treatment;
5. ECOG of 0-2;
6. Life expectancy>3 months;
7. Within 7 days (including 7 days) before screening, the laboratory test data requirements: neutrophil count ≥1.5×10^9/L, platelet count ≥90×10^9/L, hemoglobin ≥90g/L (No blood transfusion in 14 days), serum total bilirubin ≤1.25 times the upper limit of normal (ULN); ALT and AST≤2.5 x ULN (patients with liver metastases ≤5x ULN); serum creatinine ≤1.25 x ULN

Exclusion Criteria:

1. Patients who have previously been treated with albumin paclitaxel or bevacizumab or PD-1 monoclonal antibody;
2. Received any experimental drugs or anti-tumor drugs within 4 weeks prior to enrollment;
3. A history of other tumors in the past 5 years, except for cervix or basal cell carcinoma of the skin that has been cured;
4. Symptomatic brain or meningeal metastases (unless the patient receives treatment for> 6 months, the imaging results are negative within 4 weeks before entering the study, and the clinical symptoms related to the tumor are stable at the time of entering the study).

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-05-13 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-05-03 (Estimated)

PRIMARY OUTCOMES:
objective response rate (ORR) was assessed using RECIST1.1 and IRECIST standards. | Approximately 24 months
  ORR is defined as CR+PR

CONTACTS AND LOCATIONS:
Overall Officials: Xichun Hu, MD, PhD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China